CLINICAL TRIAL: NCT02570100
Title: Research and Analysis of the Mechanisms Involved in the Emergence of Breast Cancer Stem Cells
Brief Title: Research and Analysis of the Mechanisms Involved in the Emergence of Breast Cancer Stem Cells (RepriM)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The failures of the culture and immunostaining techniques for ALDH do not allow the main objective of the study to be met.
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut pour la Recherche sur le Cancer de Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RepriM-1407
Record Dates: First submitted 2015-09-29; First posted 2015-10-07 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: Cancer Stem Cells
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biological collection (Experimental): Before, during and after their treatment by chemotherapy, patients will undergo laboratory examinations.
  Interventions: Procedure: Biological collection

INTERVENTIONS:
Procedure: Biological collection — Collection of blood samples and tumor specimens :
  Biological collection before treatment :
  * 1 tumor specimen (under echographic control)
  * 4 blood collections
  Biological collection during treatment :
  * 1 tumor specimen after 3 cycles
  * 4 blood collections after 3 and 6 cycles

SUMMARY:
From a cellular perspective, breast cancers appear to develop hierarchically from a small contingent of cancer stem cells (CSCs). The presence of CSCs in tumor tissue is associated with an increased risk of recurrence and metastasis, as well as a worse prognosis. Thus, these CSCs exhibit resistance to conventional anti-tumor treatments such as radiotherapy and chemotherapy. Moreover, these treatments would favor the emergence of these CSCs and the reprogramming of non-CSCs in CSCs. It has been demonstrated in neoadjuvant that the proportion of CSCs before any treatment is correlated with chemoresistance and that a resurgence of CSCs after chemotherapy is correlated with a poor prognosis. However, the mechanisms involved in the emergence of CSCs by reprogramming of non-CSCs are not yet known.

The Oscar Lambret Center proposes a monocentric prospective interventional study based on the cellular and molecular analysis of the tumor, serum and circulating cells, before, during and at the end of the treatment for each patient receiving a neoadjuvant chemotherapy for breast cancer. The identification of the mechanisms contributing to the enrichment of CSCs resistant to chemotherapy could lead to therapeutic solutions.

DETAILED DESCRIPTION:
Patients responding criteria for selection will sign an informed consent form.

Before the initiation of chemotherapy, a tumor specimen (under echographic control) and four blood samples will be collected. The chemotherapy consists of 3 cycles of (F)EC100 spaced 21 days apart :

* Epirubicin, 100 mg/m² in intravenous (IV)
* Cyclophosphamide, 500 mg/m² in IV
* +/- 5-fluorouracile (5FU), 500 mg/m² in IV

Followed by 3 cycles of Taxotere (Docetaxel, IV, 100 mg/m²) spaced 21 days apart +/- Herceptin (Trastuzumab, IV, 8 mg/kg during C1 and then 6 mg/kg) for 1 year in the case of overexpression of the HER-2 oncoprotein.

After 3 cycles of chemotherapy (that is to say at the end of the (F)EC100 treatment, at the time of the usual ultrasound examination), a tumor specimen and four blood samples will be taken. After 6 cycles of chemotherapy (that is to say at the end of the Docetaxel +/- Trastuzumab treatment), four blood samples will be collected. A partial or total mastectomy could be performed during the 6 cycles of chemotherapy. During surgery, a tumor specimen will be taken. The indication of breast surgery will remain at the discretion of the pluridisciplinary committee of the participating center.

Prior to the start of treatment, patients will have a clinical and a paraclinical examination and will undergo laboratory examinations. On day 1 of the fourth cycle and after the sixth cycle of chemotherapy, patients will have a clinical examination and will undergo laboratory examinations. After three cycles of chemotherapy, at the time of the intermediate breast ultrasound, patients will have paraclinical examinations. Finally, at the end of the study (after partial or total mastectomy), anatomopathological examinations will be performed on the operative specimen.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18
* With a mammary adenocarcinoma histologically proven
* Who cannot benefit from a first-conserving surgery or with aggressiveness criteria on the initial biopsy (triple negative tumor, grade III histoprognostic, high Ki67, HER2 overexpressed) after presentation in multidisciplinary meeting.
* Absence of prior chemotherapy.
* Requiring a neoadjuvant chemotherapy with anthracyclines and taxanes selected in multidisciplinary meeting.
* Informed consent signed by the patient before the implementation of any specific procedure to the study.

Exclusion Criteria:

* Metastatic disease. The extension work-up is carried out according to the reference system of the participating center.
* Other histological type.
* Patient refusing the conservation of samples.
* Patient included in a clinical trial protocol with an experimental molecule (during this study).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-04; Primary Completion 2017-07 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Complete histopathological response | 1 month after surgery
  Complete histopathological response as classified by Sataloff according to the rate of CSCs before treatment.

SECONDARY OUTCOMES:
Evaluation of the expression of genes involved in reprogramming by immunohistochemistry and Reverse Transcription Polymerase Chain Reaction (RT-PCR) according to the rate of CSCs before, during and after chemotherapy. | Baseline
Evaluation of the expression of genes involved in reprogramming by immunohistochemistry and Reverse Transcription Polymerase Chain Reaction (RT-PCR) according to the rate of CSCs before, during and after chemotherapy. | After 3 cycles (cycle length = 21 days) of chemotherapy
Evaluation of the expression of genes involved in reprogramming by immunohistochemistry and Reverse Transcription Polymerase Chain Reaction (RT-PCR) according to the rate of CSCs before, during and after chemotherapy. | Within a month after surgery
Evaluation of relapse-free survival | 1 month after surgery
  Evaluation of relapse-free survival, defined as the elapsed time between the date of diagnosis and the date of appearance of a local or distant recurrence.
Quantification of the frequency of Cancer Stem Cells (CSCs) among the population of Circulating Tumor Cells (CTCs). | Baseline
Quantification of the frequency of Cancer Stem Cells (CSCs) among the population of Circulating Tumor Cells (CTCs). | After 3 cycles (cycle length = 21 days) of chemotherapy
Quantification of the frequency of Cancer Stem Cells (CSCs) among the population of Circulating Tumor Cells (CTCs). | After 6 cycles (cycle length = 21 days) of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine LAURIDANT, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No